CLINICAL TRIAL: NCT04697225
Title: Healthy Weight at Home: A Pilot Weight Loss Program for Parents of Children With a Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Towson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1181
Record Dates: First submitted 2020-12-22; First posted 2021-01-06 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- weight loss program (Experimental)
  Interventions: Behavioral: weight loss strategies; Behavioral: weight loss coaching sessions and email support

INTERVENTIONS:
Behavioral: weight loss strategies — Participants will receive recommendations on how to increase physical activity, decrease caloric intake, monitor their weight, and track the related behaviors and progress.
Behavioral: weight loss coaching sessions and email support — Participants will receive weekly coaching sessions and tailored support emails.

SUMMARY:
The objective of this study is to design, implement, and pilot a lifestyle-based, 12-week, weight loss program for parents of children with a disability. This weight loss program supports weight loss among parents. It is a first step towards a parent-only approach to promote healthier weight among children with a disability.

ELIGIBILITY:
Inclusion Criteria:

Parent

* age ≥18
* English speaking
* completion of screening and baseline data collection
* BMI ≥ 25 and weight < 300lbs (weight limit due to scale limitations)
* willing to lose weight through physical activity, weight tracking and decreased caloric intake
* willing to make changes at home to facilitate a healthy weight
* willing to complete 12 weekly weight loss video coaching sessions (20 minutes/session)
* willing to use Skype, FaceTime, Zoom, or WebEx for regular intervention contact
* Internet/ cellular plan that is sufficient for weekly program video conferencing
* willing to use the study scale with cellular technology to report weights at baseline, 12 weeks, and 24 weeks.
* willing to use the study scale with cellular technology at least weekly during the study (12 weeks)
* completion of screening and baseline data collection

Child

* age 8-18
* has a disability
* assent is required if the child is capable and willing to have height and weight taken by the parent at baseline, 12 weeks, and 24 weeks.

Exclusion Criteria:

* parent or child: previously diagnosed eating disorder, or treatment for an eating disorder
* parent: currently pregnant or plan to get pregnant in the next 6 months
* parent: planned weight loss surgery or procedure in the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Weight change among the parents at week 12 | baseline and 12 weeks
  Examine weight change (12 week - baseline) in kilograms (kg) among the parents in the 12-week weight loss program.

SECONDARY OUTCOMES:
Adherence with the scheduled weekly coaching calls | baseline to 12 weeks
  Examine the parent's adherence with the weekly coaching sessions using descriptive statistics, including percent, of coaching sessions attended.
Weight change among the parents at week 24 | baseline and 24 weeks
  Examine weight change in kg (24 week - baseline) among the parents 12 weeks after the end of the weight loss program.
Change in BMI z-score among the children | baseline, 12, and 24 weeks
  Examine changes (12 week - baseline and 24 week - baseline) in BMI-z score among the children.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Jerome, PhD, Principal Investigator — Towson University
Locations (1):
- Towson University, Towson, Maryland, United States

IPD SHARING:
Plan to Share IPD: No